CLINICAL TRIAL: NCT01723605
Title: Insitu Repair Versus Uterine Exeriorization During Cesarean Section: A Randomised Controlled Trial
Brief Title: Insitu Repair Versus Uterine Exeriorization During Cesarean Section
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Waleed El-khayat, Assisstant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 32012
Record Dates: First submitted 2012-11-04; First posted 2012-11-08 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Complications; Cesarean Section
Keywords: insitu repair; intestinal motility

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- insitu repair (Experimental): insitu repair of the uterine incision during caeserean section
  Interventions: Procedure: insitu repair
- exteriorisation of the uretus (Active Comparator): uterine closure during caeserian section with exteriorisation of the uterus
  Interventions: Procedure: exteriorisation of the uterus

INTERVENTIONS:
Procedure: insitu repair — closure of the uterine incision while the uterus initu
  Other Names: repair insitu
  Arms: insitu repair
Procedure: exteriorisation of the uterus — uterine closure while the uterus is exteriorised
  Other Names: uterine closure with exteriorisation of the uterus
  Arms: exteriorisation of the uretus

SUMMARY:
Two types of uterine repair described during cesarean section, the investigators will try to compare between the two techniques.

DETAILED DESCRIPTION:
Insitu repair of the uterus during cesarean section in Comparison to exteriorisation of the uterus during uterine closure

ELIGIBILITY:
Inclusion Criteria:

* pregnant women

Exclusion Criteria:

* liver disease
* kidney disease
* bleeding tendency
* abnormal placentation
* preeclampsia

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1000 (Actual)
Dates: Start 2012-10; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Bowel movement | 12 hours
  Regain of bowel movement

SECONDARY OUTCOMES:
Surgery duration | 2 hours
  The duration of intraoperative surgey

CONTACTS AND LOCATIONS:
Overall Officials: Waleed El-khayat, Study Chair — Cairo University
Locations (1):
- Faculty of medicine, Cairo, Egypt

REFERENCES:
- [Derived] El-Khayat W, Elsharkawi M, Hassan A. A randomized controlled trial of uterine exteriorization versus in situ repair of the uterine incision during cesarean delivery. Int J Gynaecol Obstet. 2014 Nov;127(2):163-6. doi: 10.1016/j.ijgo.2014.05.004. Epub 2014 Jun 19. PMID 25005057